CLINICAL TRIAL: NCT05406557
Title: Outcome Comparing Partial and Miniature Pulpotomy in Mature Permanent Molars With Symptomatic Partial Irreversible Pulpitis
Brief Title: Partial Versus Miniature Pulpotomy in Teeth With Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR. A RAMANI
Record Dates: First submitted 2022-05-29; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Pulpitis - Irreversible
Keywords: Irreversible pulpitis; Partial pulpotomy; Miniature pulpotomy; Vital pulp therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial pulpotomy (Active Comparator): Removal of superficial 2-3 mm of pulp tissue from entire pulp chamber
  Interventions: Procedure: Partial pulpotomy
- Miniature pulpotomy (Active Comparator): Removal of superficial 2-3 mm of pulp tissue from only affected pulp horn
  Interventions: Procedure: Miniature pulpotomy

INTERVENTIONS:
Procedure: Partial pulpotomy — In case of partial pulpotomy procedure the exposed pulp tissue will be amputated using a sterile bur in the high speed hand piece with water coolant to a depth of superficial 2-3 mm of pulp chamber.
  Arms: Partial pulpotomy
Procedure: Miniature pulpotomy — In case of miniature pulpotomy procedure the exposed pulp tissue will be amputated using a sterile bur in the high speed hand piece with water coolant to a depth of superficial 2-3 mm of only affected pulp horn
  Arms: Miniature pulpotomy

SUMMARY:
This study will compare the outcome of partial and miniature pulpotomy in mature permanent molars with symptomatic partial irreversible pulpitis

DETAILED DESCRIPTION:
After thorough history and clinical and radiographic examination, and confirmation of eligibility for the study, written informed consent will be obtained from study participants after explaining the procedure and its associated risks and benefits. Clinical diagnosis of symptomatic partial irreversible pulpitis will be established based on a history of spontaneous pain or pain exacerbated by cold stimuli and lasting for a few seconds to several hours (lingering pain) compared to control teeth and which is reproducible using cold testing.

Once included, study subjects will be randomly allocated to either Miniature Pulpotomy group or Partial Pulpotomy group. MTA (Mineral Trioxide Aggregate) will be used as pulpotomy agent. A layer of resin modified Glass Ionomer liner will be placed over the MTA and tooth will be permanently restored with composite resin in same appointment.

Pain analysis will be carried out preoperatively and postoperatively at every 24 hours till 7 days after intervention. All the subjects will be followed up for evaluation of clinical and radiographic success at 6 and 12 months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* The patient with18 -45 years of age.
* Restorable molar teeth.
* Tooth should give positive response to pulp sensibility testing.
* Clinical diagnosis of symptomatic partial irreversible pulpitis.
* Tooth with probing pocket depth and mobility are within normal limits.
* No signs of pulpal necrosis including sinus tract or swelling.
* Non-contributory medical history

Exclusion Criteria:

* Teeth with immature roots.
* No pulp exposure after caries excavation.
* Bleeding could not be controlled in 6 minutes.
* Insufficient bleeding after pulp exposure, the pulp is judged necrotic or partially necrotic

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success | Baseline to 12 Months
  Absence of spontaneous pain, discomfort, swelling, sinus tract or tenderness to palpation or percussion.
  RADIOGRAPHIC SUCCESS CRITERIA:
  No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis.
  Periapical Index score 1 or 2 according to Orstavic et al. Evaluation of both clinical and radiographic outcome is must for analyzing the actual success of therapeutic technique.
  Number of participants fulfilling both clinical as well as radiographic success criteria will be considered in success category.

SECONDARY OUTCOMES:
Pain analysis | Baseline to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain
Pulp sensibility testing | Baseline to 12 months
  To assess pulp tissue response using cold and electric pulp test at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: DR. ANKITA RAMANI, MDS, Principal Investigator — PGIDS, ROHTAK, HARYANA, INDIA-124001
Locations (1):
- Dr. Ankita Ramani, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramani A, Sangwan P, Duhan J, Popat S, Sangwan A. Effect of lateral extent of pulp tissue removal on the outcome of partial pulpotomy for managing cariously exposed mature permanent molars with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2025 Jan;58(1):71-83. doi: 10.1111/iej.14152. Epub 2024 Oct 1. PMID 39352296